CLINICAL TRIAL: NCT03957018
Title: Temporal Profile of Biomarkers Associated to Perioperative Stress Due to Carotid Endarterectomy Under Regional Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Tihamér Molnár, associate professor, University of Pecs
Other Study IDs: 4820-PTE
Record Dates: First submitted 2019-05-16; First posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Perioperative Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Carotid endarterectomy (CEA) is a high risk surgical and anesthesiological procedure. It is an essential part of stroke-prevention strategies, however the incidence of CEA related peri-operative stroke is between 5% and 10%. These procedures can be performed either in general or regional anaesthesia. We hypothesized that an appropriate awake sedation is able to decrease patient's distress and an improved satisfaction can be reached.

DETAILED DESCRIPTION:
We aim to explore the stress response of patients randomized according to different sedation protocols: (i) per os premedication only with alprazolam (BDZ group) or (ii) premedication with alprazolam combined with target control infusion (TCI) of propofol (BDZ+TCI) for awake carotid endarterectomy. A total of 50 consecutive patients with significant carotid artery stenosis will be enrolled into this prospective randomised study. All surgeries will be performed in regional anaesthesia. As premedication, all patients took 0.25 mg alprazolam 30 minutes before the procedure. After randomization 25 patients will be grouped to both arms of the study: either to "sedation with target controlled propofol infusion", or to "only premedication". Stress markers, such as cortisol plasma levels will be serially analysed: prior to surgery (T1), before (T2) and after release of carotid clamp (T3), at 2 (T4) and 24 post-operative hours (T5). Alprazolam levels were also measured before and after the surgery.

ELIGIBILITY:
Inclusion Criteria: patients with significant symptomatic or asymptomatic carotid stenosis scheduled for carotid endarterectomy, written informed consent -

Exclusion Criteria: patient declines to participate in the study

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with significant symptomatic or asymptomatic carotid stenosis scheduled for carotid endarterectomy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-11-28 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
major vascular events | at 30th postoperative day
  acute coronary syndrome, myocardial infarction, stroke, transient ischemic attack

SECONDARY OUTCOMES:
mortality and vascular events | 5-year follow-up
  death, acute coronary syndrome, myocardial infarction, stroke, transient ischemic attack

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pecs, Pécs, Baranya, Hungary